CLINICAL TRIAL: NCT01524328
Title: Complementary and Alternative Medicine in Patients With Inflammatory Bowel Disease. A Cross Sectional Study in Norway.
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/1683/
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Complementary and alternative medicine; HRQoL, Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the proportion of use of complementary and alternative medicine (CAM) in patients with inflammatory bowel disease (IBD). In addition, the reason for, and satisfaction with use of CAM.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years and with verified diagnosis of Crohn's disease or ulcerative colitis attending an outpatient clinic in a Norwegian hospital.

Exclusion Criteria:

* Patients <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with (>18 years) a verified diagnosis of Crohn's disease or ulcerative colitis attending an outpatient clinic in a Norwegian hospital.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Moum, professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Oslo County, Norway